CLINICAL TRIAL: NCT00820729
Title: The Prevalence of Pulmonary Hypertension and the Significance of Different Biomarkers in Chronic Interstitial Lung Disease
Brief Title: Biomarkers in Pulmonary Hypertension Associated to Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Charlotte Andersen, MD, University of Aarhus
Other Study IDs: Fibrosis-ECHO 2009
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Interstitial Lung Disease; Pulmonary Hypertension; Biomarkers
Keywords: interstitial lung disease; pulmonary hypertension; biomarkers; NT-pro-BNP; von Willebrand factor; D-dimer; Exhaled NO; Troponin-t
MeSH Terms: conditions — Lung Diseases, Interstitial; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with interstitial pulmonary disease

SUMMARY:
The presence of an abnormally increased pulmonary blood pressure worsens the prognosis of patients with interstitial pulmonary disease.

The aim of this study is to estimate the frequency of an increased blood pressure in the lungs among patient with interstitial pulmonary disease, and to evaluate the use of different biomarkers in diagnosis of the condition.

DETAILED DESCRIPTION:
The presence of increased pulmonary blood pressure is established by echocardiography and confirmed by right heart catheterization.

The ability of NT-proBNP, vWf, troponin-t, D-dimer and exhaled NO to predict the presence of increased pressure in the pulmonary circulation is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patients with interstitial pulmonary disease.
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Pulmonary Diseases, Århus Sygehus, Aarhus
  - Department of Cardiology, Skejby sygehus, Århus N